CLINICAL TRIAL: NCT00272870
Title: A Pilot Study of Temozolomide and 06Benzylguanine for Treatment of Newly Diagnosed High Grade Glioma, Using Autologous Peripheral Blood Stem Cells Genetically Modified for Chemoprotection
Brief Title: Treatment of Newly Diagnosed Brain Tumors With Chemotherapy and Radiation Using Cells Modified for Chemoprotection and an Experimental Drug to Decrease the Tumor Cell Resistance to Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual; drug availability
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCHMCEH003
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Glioblastoma Multiforme (WHO Grade IV); Anaplastic Astrocytoma (WHO Grade III)
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 06Benzylguanine — 120 mg/m2/day; given Day 1-5 for up to 6 courses in Block 3
Genetic: MGMT P140K — Gene manipulated cells, patients are not expected to receive greater than approximately 10 x 10e6 transduced CD34+ cells/kg
Device: Meltenyi CliniMacs — Device used for CD34+ cell separation of peripheral collection

SUMMARY:
Cure rates for patients with high grade glioma remain disappointing, in part because tumor cells are often resistant to chemotherapy, and because using higher doses of chemotherapy causes damage to normal blood cells. This trial is designed to try to overcome both of these barriers. The idea is to make tumor cells more sensitive to a chemotherapy agent, Temozolomide, by using 06Benzylguanine (06BG). In addition, patients will have a portion of their blood cells modified by the insertion of a chemotherapy resistance gene which may help protect blood cells from damage by the combination of the Temozolomide and 06BG.

DETAILED DESCRIPTION:
The use of temozolomide (TEM) both during and after irradiation is a promising new approach for the treatment of patients with high-grade glioma. However, this treatment is limited by tumor cell resistance and therapy-related hematologic toxicity. To overcome TEM resistance, in this study we will add the chemotherapy sensitizing drug O6-Benzylguanine (BG). To overcome hematologic toxicity, patients will receive autologous hematopoietic stem cells transduced with a chemotherapy resistance gene designed to protect these cells from subsequent therapy with this drug combination.

The potential benefit of using transduced blood stem cells is the possibility for dose escalation of TEM, since hematologic toxicity has heretofore limited higher doses. Transduction will be accomplished with a retroviral vector carrying MGMTP140K, which codes for a mutated form of the resistance protein methylguanine-DNA methyltransferase (MGMT). Successful transduction of hematopoietic cells with MGMTP140K makes them resistant to the toxic effects of both TEM + BG. Repeated doses of these drugs should therefore result in an increase in the percentage of transduced (and thus protected) blood stem cells, thus reducing the likelihood of hematologic toxicity with further therapy. Accordingly, patients who are tolerating therapy well and who have laboratory evidence of chemoprotection will receive intrapatient dose escalation of TEM + BG during courses 2-6.

Eligible patients must be between 5 and 55 years of age and have newly-diagnosed high-grade glioma (anaplastic astrocytoma or glioblastoma multiforme) which cannot be completely resected. No prior therapy other than surgery is allowed, and patients must have adequate performance status and organ function as defined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Age > 5 years and < 55 years. NOTE: Subjects ages 5-30 are eligible to be treated at Cincinnati Children's Hospital Medical Center; subjects over age 30 will be treated at Ohio State University Comprehensive Cancer Center.

3.1.2 Anticipated life expectancy of at least nine months 3.1.3 Karnofsky score > 50 for patients > 10 years of age, and Lansky score > 50 for patients < 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

3.1.4 Patients must have one of the following newly-diagnosed central nervous system tumors, confirmed by histologic verification: Glioblastoma multiforme (WHO grade IV) OR Anaplastic astrocytoma (WHO grade III)

3.1.5 Patients older than 30 years that have undergone a gross total resection and who do not have measurable disease on post operative MRI; measurable disease as assessed by post operative MRI is required on patients 30 years of age or younger.

3.1.6 Neurologic deficits and corticosteroid doses must be stable or decreasing at the time of study entry.

3.1.7 Adequate organ function as defined by: Serum creatinine < upper limit of normal, or GFR > 70 ml/min/1.73 m2 Total bilirubin < 2.0 mg/dl; SGPT (ALT) AND SGOT (AST) < 2.5x upper limit of normal; serum albumin > 2.0 g/dL Absolute neutrophil count > 1,000/µl, platelet count > 75,000/µl independent of transfusions

3.1.8 The patient and/or the patient's legally authorized guardian must give written informed consent according to local Institutional and/or University Human Experimentation Committee requirements.

3.1.9 Women or men with reproductive potential must use effective contraception throughout the study. Effective contraception methods for women would include either an oral or transdermal contraceptive, injectable contraceptive (e.g., Depo-Provera), or contraceptive implants (e.g., intrauterine device). All males on study must agree to the use of condoms during intercourse.

3.1.10 Women of reproductive potential must have a negative serum pregnancy test.

Exclusion Criteria:

3.2.1 Any prior treatment with chemotherapy or radiotherapy.

3.2.2 Any tumor arising in the spine or brainstem.

3.2.3 Presence of metastatic disease in the spine.

3.2.4 WHO grade III oligodendroglioma or oligoastrocytoma.

3.2.5 Active infection at time of study entry.

3.2.6 Pregnant or lactating females are excluded, because of the known teratogenic effects of alkylating agents.

3.2.7 Known HIV-positive patients. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy and are excluded from this study. An infectious disease screen consisting of HIV I & II Ab and NAT, HTLV I & II Ab, RPR, Hepatitis B Surface Ag, Hepatitis B Core Ab and Hepatitis C Ab will be obtained at study entry.

3.2.8 Concurrent treatment with other investigational anti-cancer agents.

3.2.9 Serious illness or medical condition which would not permit the patient to be managed according to the protocol.

3.2.10 Low-grade glioma (WHO Grade 1-2).

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and feasibility of infusing autologous PBSC transduced with MSCV-MGMTP140K construct, using the fibronectin component CH-296 to assist gene transfer. | 5 years

SECONDARY OUTCOMES:
Assess the efficiency of gene transfer and durability of transgene expression in this clinical setting. | 5 years
Assess the degree of chemotherapy resistance in transduced cells, and the ability to enrich the population of transduced stem cells with subsequent courses of chemotherapy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Punam Malik, MD, Study Director — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States